CLINICAL TRIAL: NCT06015373
Title: The Impact of Carvedilol Posology on Clinically Significant Portal Hypertension: Insights From Elastography Measurements
Brief Title: The Impact of Carvedilol Posology on Clinically Significant Portal Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar De São João, E.P.E. (Other)
Responsible Party: Principal Investigator, Bruno Besteiro, MD, Principal Investigator, Centro Hospitalar De São João, E.P.E.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LHU-2023-001
Record Dates: First submitted 2023-08-11; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Clinically Significant Portal Hypertension
Keywords: portal hypertension; carvedilol; elastography
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with CSPH receiving carvedilol twice daily and supress the night dose of carvedilol (Experimental): In this experimental study, 34 patients with CSPH receiving carvedilol twice daily were asked to supress the night dose of carvedilol, in order to have a dose interval of approximately 24 hours. Spleen stiffness measurement (SSM) by transient elastography (TE) was performed and compared with SSM prior or under treatment. Same procedure was applied to liver stiffness measurement (LSM).
  Interventions: Drug: supress the night dose of carvedilol

INTERVENTIONS:
Drug: supress the night dose of carvedilol — already described

SUMMARY:
Carvedilol has emerged as the preferred non-selective β-blocker (NSBB) for treating portal hypertension. However, there is still a debate in dosing regimen, specially regarding dose interval, with a potential lower bioavalability in once daily regimens. The aim of this study is to assess the acute effects of carvedilol posology in patients with clinically significant portal hypertension (CSPH), as a surrogate marker of bioavailability.

In this experimental study, patients with CSPH receiving carvedilol twice daily were asked to supress the night dose of carvedilol, in order to have a dose interval of approximately 24 hours. Spleen stiffness measurement (SSM) by transient elastography (TE) was performed and compared with SSM prior or under treatment. Same procedure was applied to liver stiffness measurement (LSM).

ELIGIBILITY:
Inclusion Criteria:

* patients with CSPH (defined as a LSM 25 kPa or SSM over 45kPa prior to introduction of carvedilol)

Exclusion Criteria:

* Non-responders to non-selective β-blockers (NSBB)
* NSBB other than carvedilol
* Dosing regimen other than twice daily
* No SSM or LSM within 3 months prior to the beginning of the study
* Body mass index (BMI) > 30 m/kg2
* Contraindications to NSBB use
* Portal venous thrombosis
* Refusal to participate in the study
* Failure to comply to the study regimen

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
spleen stiffness measurement (SSM) | Baseline SSM measured up to 3 months before enrolment, and measured at 24 hours after suspending carvedilol
  Change from baseline in spleen stiffness measurement (SSM) measured by transient elastography (TE) after 24 hour suspension of carvedilol treatment.

SECONDARY OUTCOMES:
liver stiffness measurement (LSM) | Baseline LSM measured up to 3 months before enrolment, and measured at 24 hours after suspending carvedilol
  Change from baseline in liver stiffness measurement (LSM) measured by transient elastography (TE) after 24 hour suspension of carvedilol treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar de Trás os Montes e Alto Douro, Vila Real, Lordelo, Portugal

DOCUMENTS (2):
  • Study Protocol (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT06015373/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT06015373/SAP_001.pdf